CLINICAL TRIAL: NCT02546570
Title: Posttraumatic Stress Disorder and Affective Functioning: A Test of the Potentially Normalizing Effects of Oxytocin
Brief Title: Oxytocin and Affect Processing in Posttraumatic Stress Disorder
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Center for PTSD (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1502015347
Record Dates: First submitted 2015-06-15; First posted 2015-09-11 (Estimated); Results first posted 2020-04-08 (Actual); Last update posted 2020-04-08 (Actual); Status verified 2020-03

CONDITIONS: Posttraumatic Stress Disorder (PTSD)
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Oxytocin; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Healthy adult controls (18-55) (Experimental): Drug: oxytocin and placebo nasal spray (within-subjects design, blinded and counterbalanced for two lab sessions); dosage=24 international units (IU). Participant inserts nasal spray container 1cm into nostril at angle of 45 degrees and sprays. Will wait 15 seconds then repeat administration to other nostril (alternating between nostrils). Participants will receive 6 puffs in total (3 in each nostril).
  Interventions: Drug: Oxytocin; Drug: Placebo
- Adults with PTSD (18-55) (Experimental): Drug: oxytocin and placebo nasal spray (within-subjects design, blinded and counterbalanced for two lab sessions); dosage=24 international units (IU). Participant inserts nasal spray container 1cm into nostril at angle of 45 degrees and sprays. Will wait 15 seconds then repeat administration to other nostril (alternating between nostrils). Participants will receive 6 puffs in total (3 in each nostril).
  Interventions: Drug: Oxytocin; Drug: Placebo
- Trauma-exposed/no-PTSD adults (18-55) (Experimental): Drug: oxytocin and placebo nasal spray (within-subjects design, blinded and counterbalanced for two lab sessions); dosage=24 international units (IU). Participant inserts nasal spray container 1cm into nostril at angle of 45 degrees and sprays. Will wait 15 seconds then repeat administration to other nostril (alternating between nostrils). Participants will receive 6 puffs in total (3 in each nostril).
  Interventions: Drug: Oxytocin; Drug: Placebo

INTERVENTIONS:
Drug: Oxytocin — See arm/group descriptions for dosage amount and procedure.
  Other Names: Pitocin
Drug: Placebo — See arm/group descriptions for dosage amount and procedure.
  Other Names: saline

SUMMARY:
The investigators will use multiple methods (including Oxytocin intranasal inhalation, neuroimaging, behavioral measures, peripheral hormone measurements) to examine how individuals' behavior, cognition, and brain function is impacted by the neuro-hormone Oxytocin. Specifically, the investigators plan to evaluate the influence of Oxytocin administration on affective processing in non-trauma exposed and trauma-exposed adults (both with and without posttraumatic stress disorder, PTSD).

DETAILED DESCRIPTION:
The investigators will use multiple methods (including Oxytocin intranasal inhalation, neuroimaging, behavioral measures, peripheral hormone measurements) to examine how individuals' behavior, cognition, and brain function is impacted by the neuro-hormone Oxytocin. Specifically, the investigators plan to evaluate the influence of Oxytocin administration on affective processing in non-trauma exposed and trauma-exposed adults (both with and without posttraumatic stress disorder, PTSD). The investigators expect oxytocin (compared to placebo) to positively influence affect processing in healthy subjects, as well as among those diagnosed with PTSD. Given current literature, the investigators expect oxytocin to elevate the processing\perception of positive-related stimuli, and reduce the salience of aversive or un-pleasant cues. The investigators expect oxytocin to impact participants' brain function as measured with functional magnetic resonance imaging (fMRI) while visually processing social and affect-related stimuli, rendering brain function and affective processing to be "more typical" or "adaptive" compared to placebo. Oxytocin's effect on human repertoire is not necessarily direct, but can interact with the individual's socioemotional characteristics, early life environment, and psychiatric symptoms. Therefore, the investigators will incorporate measures that capture the various dimensions that likely shape the effect of oxytocin.

ELIGIBILITY:
Inclusion Criteria:

* Adults: age 18-55
* Be in good medical health
* Be cooperative with testing
* English is a language spoken in the family
* PTSD as diagnosed by a certified clinician or the research team for PTSD group.

Exclusion Criteria:

* Moderate or severe acute or chronic medical illnesses (e.g.cardiac disease, diabetes, epilepsy, influenza).
* History of hypertension with baseline blood pressure above 160 mm Hg (systolic) over 100 mm Hg (diastolic).
* history of syncope and/or baseline blood pressure below 100 mm Hg (systolic).
* weight >300lb
* The use of some psychotropic medications will not be allowed. Females taking contraceptive hormones will not be able to participate in the study.
* Currently breast feeding or pregnant
* For MRI ONLY: Any metal or electromagnetic implants
* For MRI ONLY: Significant hearing loss or other severe sensory impairment
* A fragile health status.
* For MRI ONLY: A history of seizures or current use of anticonvulsants
* Healthy adult controls (HC):
* Be free of both neurological and psychiatric disorders (current and past) on the basis of self-report
* Be free of psychiatric disorders

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 11 (Actual)
Dates: Start 2015-08 (Actual); Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Linda Mayes, MD, Principal Investigator — Yale University
Locations (1):
- Yale University, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Groups:
- Adults With PTSD (18-55); Trauma-exposed/No-PTSD Adults (18-55): Drug: oxytocin and placebo nasal spray (within-subjects design, blinded and counterbalanced for two lab sessions); dosage=24 international units (IU). Participant inserts nasal spray container 1cm into nostril at angle of 45 degrees and sprays. Will wait 15 seconds then repeat administration to other nostril (alternating between nostrils). Participants will receive 6 puffs in total (3 in each nostril).
  Oxytocin: See arm/group descriptions for dosage amount and procedure. Placebo: See arm/group descriptions for dosage amount and procedure.
Period: Overall Study
Arm/Group | Adults With PTSD (18-55) | Trauma-exposed/No-PTSD Adults (18-55)
Started | 9 | 2
Crossover Order: Oxytocin, Placebo | 6 | 2
Crossover Order: Placebo, Oxytocin | 3 | 0
Completed | 9 | 2
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Combat Veterans
Groups:
- Total: Total of all reporting groups
Arm/Group | Adults With PTSD (18-55) | Trauma-exposed/No-PTSD Adults (18-55) | Total
Number analyzed (Participants) | 9 | 2 | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 9 | 2 | 11
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 9 | 2 | 11

OUTCOME MEASURES:

1. Primary Outcome: fMRI Analysis: Change in Anterior Insula Region
Description: Change in blood-oxygen-level dependent (BOLD) contrast signal in regions of interest relevant to fear/threat (e.g., decrease in amygdala activation) and reward processing (increase in ventral striatum activation) in oxytocin versus placebo sessions.
  Forearm brush stroking targets C-tactile (CT) nerves, which respond to gentle touch and engage the insula and cortical brain regions that mediate social-emotional processing. Palm brush stroking is the control condition, in that CT afferents do not innervate the palm. We contrasted BOLD responses to gentle continuous brushing of the arm vs. palm (4 blocks of 8 trials each), expecting greater oxytocin-related increases in brain reactivity within the insula and other regions in the forearm condition versus the palm condition. The values are % signal change from baseline.
Time Frame: 1 week; fMRI data collected at second and third visits, one week apart
Population: Data for all enrolled are summarized.
Measure: Mean (95% Confidence Interval); unit: percentage of area activation
Groups:
- Adults With PTSD (18-55): Drug; Adults With PTSD (18-55): Placebo; Adults Without PTSD (18-55): Drug; Adults Without PTSD (18-55): Placebo: Drug: oxytocin and placebo nasal spray (within-subjects design, blinded and counterbalanced for two lab sessions); dosage=24 international units (IU). Participant inserts nasal spray container 1cm into nostril at angle of 45 degrees and sprays. Will wait 15 seconds then repeat administration to other nostril (alternating between nostrils). Participants will receive 6 puffs in total (3 in each nostril).
  Oxytocin: See arm/group descriptions for dosage amount and procedure.
  Placebo: See arm/group descriptions for dosage amount and procedure.
Arm/Group | Adults With PTSD (18-55): Drug | Adults With PTSD (18-55): Placebo | Adults Without PTSD (18-55): Drug | Adults Without PTSD (18-55): Placebo
Number analyzed (Participants) | 9 | 9 | 2 | 2
percentage of area activation
  forearm | -12.6 [-39.7 to 14.3] | -1.6 [-13.5 to 10.3] | 10.6 [-100 to 100] | -7.8 [-64.4 to 48.8]
  palm | -13.9 [-39.7 to 11.8] | 3.9 [-12.9 to 20.9] | 5.9 [-100 to 100] | 3.6 [-100 to 100]

2. Primary Outcome: fMRI Analysis: Change in Accumbens Region
Description: as for outcome 1
Time Frame: 1 week; fMRI data collected at second and third visits, one week apart
Population: Data for all enrolled are summarized.
Measure: Mean (95% Confidence Interval); unit: percentage of area activation
Arm/Group | Adults With PTSD (18-55): Drug | Adults With PTSD (18-55): Placebo | Adults Without PTSD (18-55): Drug | Adults Without PTSD (18-55): Placebo
Number analyzed (Participants) | 9 | 9 | 2 | 2
percentage of area activation
  forearm | 7.6 [-5.4 to 20.7] | -7.9 [-17.3 to 1.5] | -17.2 [-100 to 100] | -12.7 [-70.6 to 45.1]
  palm | -14.8 [-25.8 to -3.9] | -8.0 [-25.4 to 9.3] | -8.5 [-87.8 to 70.7] | 1.2 [-100 to 100]

3. Primary Outcome: fMRI Analysis: Change in Amygdala Region
Description: as for outcome 1
Time Frame: 1 week; fMRI data collected at second and third visits, one week apart
Population: Data for all enrolled are summarized.
Measure: Mean (95% Confidence Interval); unit: percentage of area activation
Arm/Group | Adults With PTSD (18-55): Drug | Adults With PTSD (18-55): Placebo | Adults Without PTSD (18-55): Drug | Adults Without PTSD (18-55): Placebo
Number analyzed (Participants) | 9 | 9 | 2 | 2
percentage of area activation
  forearm | -3.8 [-13.7 to 6.1] | -9.1 [-20.6 to 2.3] | 14.5 [-24.9 to 54.1] | -6.7 [-74.8 to 61.3]
  palm | -4.2 [-13.6 to 5.2] | .58 [-11.0 to 12.2] | 16.7 [-100 to 100] | -.45 [-90.2 to 89.4]

4. Primary Outcome: fMRI Analysis: Change in dACC Region
Description: as for outcome 1
Time Frame: 1 week; fMRI data collected at second and third visits, one week apart
Population: Data for all enrolled are summarized.
Measure: Mean (95% Confidence Interval); unit: percentage of area activation
Groups:
- Adults With and Without PTSD (18-55): Drug; Adults With and Without PTSD (18-55): Placebo; Adults Without PTSD (18-55): Drug; Adults Without PTSD (18-55): Placebo: Drug: oxytocin and placebo nasal spray (within-subjects design, blinded and counterbalanced for two lab sessions); dosage=24 international units (IU). Participant inserts nasal spray container 1cm into nostril at angle of 45 degrees and sprays. Will wait 15 seconds then repeat administration to other nostril (alternating between nostrils). Participants will receive 6 puffs in total (3 in each nostril).
  Oxytocin: See arm/group descriptions for dosage amount and procedure.
  Placebo: See arm/group descriptions for dosage amount and procedure.
Arm/Group | Adults With and Without PTSD (18-55): Drug | Adults With and Without PTSD (18-55): Placebo | Adults Without PTSD (18-55): Drug | Adults Without PTSD (18-55): Placebo
Number analyzed (Participants) | 9 | 9 | 2 | 2
percentage of area activation
  forearm | -20.9 [-52.6 to 10.7] | -16.4 [-28.2 to -4.6] | -4.8 [-6.6 to -3.0] | -30.2 [-62.3 to 1.8]
  palm | -23.8 [-48.3 to 0.5] | -7.5 [-25.0 to 9.9] | -10.9 [-100 to 100] | -12.7 [-65.7 to 40.3]

5. Primary Outcome: fMRI Analysis: Change in mOFC Region
Description: as for outcome 1
Time Frame: 1 week; fMRI data collected at second and third visits, one week apart
Population: Data for all enrolled are summarized.
Measure: Mean (95% Confidence Interval); unit: percentage of area activation
Arm/Group | Adults With PTSD (18-55): Drug | Adults With PTSD (18-55): Placebo | Adults Without PTSD (18-55): Drug | Adults Without PTSD (18-55): Placebo
Number analyzed (Participants) | 9 | 9 | 2 | 2
percentage of area activation
  forearm | 1.5 [-6.8 to 9.8] | 2.5 [-6.8 to 22.7] | 1.7 [-92.6 to 96.2] | -8.1 [-100 to 100]
  palm | -4.9 [-18.2 to 8.2] | 12.3 [2.0 to 22.7] | 4.2 [-46.3 to 54.9] | 10.3 [-21.6 to 23.7]

6. Primary Outcome: fMRI Analysis: Change in rACC Region
Description: as for outcome 1
Time Frame: 1 week; fMRI data collected at second and third visits, one week apart
Population: Data for all enrolled are summarized.
Measure: Mean (95% Confidence Interval); unit: percentage of area activation
Arm/Group | Adults With PTSD (18-55): Drug | Adults With PTSD (18-55): Placebo | Adults Without PTSD (18-55): Drug | Adults Without PTSD (18-55): Placebo
Number analyzed (Participants) | 9 | 9 | 2 | 2
percentage of area activation
  forearm | -5.9 [-16.0 to 4.0] | -4.4 [-12.0 to 3.0] | -0.2 [-15.2 to 14.8] | -16.3 [-36.7 to 4.1]
  palm | -9.2 [-21.9 to 3.4] | 0.7 [-7.7 to 9.3] | -1.6 [-100 to 100] | -7.6 [-100 to 100]

7. Primary Outcome: fMRI Analysis: Change in vmPFC Region
Description: as for outcome 1
Time Frame: 1 week; fMRI data collected at second and third visits, one week apart
Population: Data for all enrolled are summarized.
Measure: Mean (95% Confidence Interval); unit: percentage of area activation
Arm/Group | Adults With and Without PTSD (18-55): Drug | Adults With and Without PTSD (18-55): Placebo | Adults Without PTSD (18-55): Drug | Adults Without PTSD (18-55): Placebo
Number analyzed (Participants) | 9 | 9 | 2 | 2
percentage of area activation
  forearm | -3.8 [-10.5 to 2.7] | -6.8 [-13.0 to -0.6] | -3.3 [-24.8 to 18.0] | -16.0 [-96.7 to 64.6]
  palm | -12.0 [-26.6 to 2.5] | 2.4 [-7.4 to 12.4] | -2.8 [-67.5 to 61.7] | -10.4 [-100 to 100]

8. Secondary Outcome: Salivary Oxytocin
Description: Expect within-session (30 min) increase in peripheral salivary oxytocin level during OT sessions (within-session), and higher OT levels in oxytocin administration vs. placebo sessions. Peripheral OT levels measured with Salivettes (sterile cotton participants will be asked to chew on for 1 minutes).
Time Frame: Within session (30 min) and between sessions (1 week); saliva samples collected twice (before and after OT administration) at both second and third visits, one week apart
Population: Saliva samples were collected as outlined. The research team attempted to analyze them. However, despite best efforts, and assurances from the manufacturer, the assay performance remained unacceptable primarily in regards to inadequate sensitivity and significant variability in sample duplicates. Therefore, there are no results to report.
Arm/Group | Adults With PTSD (18-55): Drug | Adults With PTSD (18-55): Placebo | Adults Without PTSD (18-55): Drug | Adults Without PTSD (18-55): Placebo
Number analyzed (Participants) | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Arm/Group | Adults With PTSD (18-55) | Trauma-exposed/No-PTSD Adults (18-55)
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/2
Other Adverse Events (participants affected / at risk) | 0/9 | 0/2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No